CLINICAL TRIAL: NCT00851851
Title: New Non-invasive Methods for Real-time Monitoring of Organ Function.
Acronym: RTMKF
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201110033
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Acute Renal Failure; Chronic Renal Failure
Keywords: Surgical patients
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Measuring novel proteins in the urine of surgical patients that can be used to diagnose impending acute or chronic renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age

Exclusion Criteria:

* Patients at end stage renal disease
* Patients dependent on dialysis at time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients.
Sampling Method: Probability Sample
Enrollment: 641 (Actual)
Dates: Start 2009-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To identify acute, chronic or lack of renal failure | Pre-op, intraoperative, post operatively (1-6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Morrissey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States